CLINICAL TRIAL: NCT06661954
Title: Sacral Interface Pressure Mapping of Hospital Bed Systems
Brief Title: Comparison of Sacral Interface Pressure in Healthy Volunteers on Two Dynamic Pressure-Prevention Support Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rachel Cowan, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300012406
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer; Pressure Distribution
Keywords: Pressure Injury; Pressure Mapping
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy Adult Volunteers (Experimental): One Arm. Repeated measures. All participants are assessed in each of the four bed-position configurations. Bed-position assessment sequence is randomized for each participant.
  Interventions: Device: Bed A - Head of Bed 0 degrees; Device: Bed B - Head of Bed 0 degrees; Device: Bed A - Head of bed at 30 degrees; Device: Bed B - head of bed at 30 degrees

INTERVENTIONS:
Device: Bed A - Head of Bed 0 degrees — Low air loss mattress in supine position
Device: Bed B - Head of Bed 0 degrees — Standard hospital mattress in supine position
Device: Bed A - Head of bed at 30 degrees — Low air loss mattress with head of bed at 30 degrees
Device: Bed B - head of bed at 30 degrees — Standard hospital mattress with head of bed at 30 degrees

SUMMARY:
The purpose of the research study is to investigate the peak sacral interface pressures of two separate hospital bed systems in the supine and 30 degrees head-of-bed elevation position.

ELIGIBILITY:
Inclusion Criteria:

* non-disabled
* can walk & stand independently
* can visit UAB SIM Lab once for 45 to 60 minutes

Exclusion Criteria:

-skin breakdown or compromising skin conditions

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Cowan, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified data set will be shared upon request contingent on execution of a data sharing/use agreement between the PI's institution and the individual/institution/organization requesting the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Convivence sample of healthy non-disabled adults were recruited from personal and professional contacts of the study team and word of mouth. Recruitment occurred from 6/11/2024 through 10/23/2024
Pre-assignment Details: The protocol did not include any events between enrollment and assignment. All enrolled participants completed the protocol
Groups:
- Healthy Adult Volunteers: One Arm. Repeated measures. All participants are assessed in each of the four bed-position configurations. Bed-position assessment sequence is randomized for each participant.
  Bed A - Low air loss mattress with head of bed at 0 degrees
  Bed B - Standard hospital mattress with head of bed at 0 degrees
  Bed A - Low air loss mattress with head of bed at 30 degrees
  Bed B - Standard hospital mattress with head of bed at 30 degrees
Period: Overall Study
Arm/Group | Healthy Adult Volunteers
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Adult Volunteers
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18
Height (inches) [Mean (Standard Deviation); unit: inches] | 67.9 (4.5)
Weight (pounds) [Mean (Standard Deviation); unit: pounds] | 171.9 (32.3)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 26.1 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Peak Sacral Pressure
Description: Peak sacral pressure is defined as the highest pressure within a 9-10 cm squared area under the coccyx. The area under coccyx was identified prior to each condition tested using the pressure mapping system. Presure was recorded continuously for 15 minutes. Because the mattresses tested were advertised as 'cycling' pressure, with the cycles set to 5 minutes, the average of minutes 1-3 and 6-8 were used for analysis. These periods represent different phases of the 'cycling' where sacral pressure would conceivably differ.
Time Frame: minutes 1-3 and minutes 6-8
Population: 18 participants completed the data collection protocol. 16 participants were included in the analysis. 2 participants were excluded from all analyses after inspection of their data suggested the position of the coccyx had been misidentified.
Measure: Mean (Standard Deviation); unit: mm hg
Arm/Group | Healthy Adult Volunteers
Number analyzed (Participants) | 16
mm hg
  Bed A, Head of Bed 0 degrees Minutes 1-3 | 17.8 (4.2)
  Bed B, Head of Bed 0 degrees Minutes 1-3 | 21.0 (4.5)
  Bed A, Head of Bed 0 degrees Minutes 6-8 | 17.1 (4.9)
  Bed B, Head of Bed 0 degrees Minutes 6-8 | 21.6 (4.6)
  Bed A, Head of Bed 30 degrees Minutes 1-3 | 17.3 (6.0)
  Bed B, Head of Bed 30 degrees Minutes 1-3 | 24.9 (8.7)
  Bed A, Head of Bed 30 degrees Minutes 6-8 | 16.9 (5.2)
  Bed B, Head of Bed 30 degrees Minutes 6-8 | 25.7 (8.6)
Statistical Analysis 1: Comparison: Healthy Adult Volunteers; Peak sacral pressure (mmHg) was collected for every minute of the 10 minute recording. Two averages for each test condition were analyzed (Minutes 1-3 (Min1-3) and 6-8 (Min6-8)). These averages capture pressure during two different 5 minute cycles, when conceivably, sacral pressure would differ. Paired t-tests compared pressure of Bed A and Bed B at each time at each head of bed position (4 tests, two-tailed test, alpha=0.05). A Holm-Bonferroni correction controlled type 1 error; Test type: Other — paired t-tests were used to identify statistically significant differences; p < 0.05, t-test, 2 sided — Paired t-tests compared pressure of Bed A and Bed B at each time at each head of bed position (4 tests, two-tailed test, alpha=0.05). A Holm-Bonferroni correction was used to control type 1 error

ADVERSE EVENTS:
Time Frame: From signing of the informed consent form until getting off the final Bed-Position that was tested. All testing occurred during one visit to the laboratory lasting up to 90 minutes.
Arm/Group | Healthy Adult Volunteers
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
The pressure mapping system used to record peak pressures was a clinical system. This system does not allow for export of the continuous recording. One minute averages had to be computed on the clinical system and then manually transcribed into excel.

Participants self-palpated the location of the ischial tuberosities and coccyx. These regions were then labelled on the clinical pressure mapping system.

These methodological limitations are assumed to decrease precision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT06661954/Prot_SAP_000.pdf